CLINICAL TRIAL: NCT00982293
Title: A Randomized, Double Blind, Placebo Controlled Study of the Application of Magnetic Fields Using the Resonator in Adjunctive Management of Type 2 Diabetes Mellitus, Pilot Study II
Brief Title: The Application of Extremely Low Level Magnetic Fields as Adjunctive Treatment for Type II Diabetes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in Recruitment
Sponsor: pico-tesla Magnetic Therapies, LLC (Industry)
Responsible Party: Allen S. Braswell CEO, pico-tesla Magnetic Therapies, LLC
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 09109-01
Record Dates: First submitted 2009-09-21; First posted 2009-09-23 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active fields (Active Comparator)
  Interventions: Device: Resonator device
- Inactive device (Sham Comparator): Placebo treated group, will receive the 3 times weekly for 13 weeks (39) sessions, however, the device will not be "on".
  Interventions: Device: Resonator device - sham

INTERVENTIONS:
Device: Resonator device — Low level electromagnetic fields for whole body immersion, 3 times weekly for 13 weeks (39) sessions of approximately 11/2 hours each.
  Arms: Active fields
Device: Resonator device - sham — Treatment, 3 times weekly for 13 weeks (39) sessions - device will not be "on"
  Arms: Inactive device

SUMMARY:
The purpose of this study is to see if using a device called the Resonator, that puts out very low level electromagnetic fields, effects blood glucose and A1c levels in people with Type 2 Diabetes.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine whether application of magnetic fields generated by the Resonator TM, as an adjunctive therapy to oral medications results in statistically significant reductions in fasting blood glucose levels, post prandial glucose levels and hemoglobin A1c levels. The study will also investigate any induced changes in serum lipids.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of Type 2 Diabetes Mellitus with a hemoglobin A1c level above 7.5%, despite management of diabetes with diet and/or medication.
* Subject currently performs routine finger stick blood sugar testing as part of his or her current diabetes disease management regimen.
* Subject is ambulatory
* Subject is on stable oral medication regimen without significant side effects for at least three (3) months (stable insulin regimen NOT permissible); willingness and ability to maintain the stable oral medication regimen throughout the course of the study. If on agents suspected of contributing to hyperglycemia(see list below), subject must have been on a stable dose of this(these) agent(s) for 6 months prior to study initiation.
* Hemoglobin A1c levels within a 0.8 % range of patient mean A1c level for the last two documented determinations, that must be within 2 years of the baseline testing date.
* Willingness to test finger stick blood sugars according to prescribed protocol.
* Willingness to have lab test blood draws performed according to prescribed protocol
* Willingness to maintain stable diet and activity regimen for the duration of the study.
* Willing and able to abstain from partaking in any non-essential (not physician ordered) existing or new treatments to improve serum blood sugar levels
* Willing and able to abstain from all medications that could affect diabetes mellitus and/or any of its associated symptoms for the duration of the study
* Adequate contraceptive measures for females subjects
* Any ethnic background

Exclusion Criteria:

* Change in medical regimen within 3 months prior to initiation of study.
* Any signs of type 1 diabetes mellitus (including any history of ketoacidosis or new requirement for insulin therapy within the 6 month period prior to study initiation).
* Active significant infectious process within 3 weeks of study initiation causing wide fluctuations in finger stick blood sugar level
* Change in BMI of greater than 6 % within a 3 month period prior to study initiation
* Any planned revascularization procedure.
* Symptomatic congestive heart failure.
* Leg or foot ulceration or open wounds
* Gangrene.
* History of intermittent claudication
* Hemodialysis
* Currently being treated for malignancy
* Currently being treated with oral or intravenous catabolic steroids
* Reported consumption of more than 14 alcoholic drinks per week.
* Pregnant, breast feeding, or planning pregnancy prior to the end of participation
* Developmental disability or cognitive impairment that would make it difficult for the subject to partake in the clinical study, including adequate comprehension of the informed consent form and ability to record the necessary measurements
* Uncontrolled hypertension
* Uncontrolled atrial fibrillation or other uncontrolled arrythmias, e.g. tachycardia, bradycardia
* Uncontrolled seizure disorder
* Uncontrolled, unstable, or untreated medical conditions which may significantly impact the subject's health or ability to complete the entire study, in the opinion of the investigator.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the improvement in Subject's hemoglobin A1c level after 13 weeks of treatment compared to baseline. | baseline, end of treatment (13 weeks) and 3 months post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- pico-tesla Magnetic Therapies, Littleton, Colorado, United States